CLINICAL TRIAL: NCT03436589
Title: Understanding the Immediate and Long-term Effects of Supplemental Nutrition Assistance Program-Education as an Intervention to Improve Food Security Among Households With Children in Indiana
Brief Title: The Indiana SNAP-Ed Long-term Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Purdue University (Other)
Collaborators: University of Kentucky Center for Poverty Research (Unknown); North Central Nutrition Education Center of Excellence (Unknown)
Responsible Party: Principal Investigator, Heather Eicher-Miller, Assistant Prof. of Nutrition Sciences, Purdue University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1306013723
Record Dates: First submitted 2018-02-12; First posted 2018-02-19 (Actual); Last update posted 2018-02-19 (Actual); Status verified 2018-02

CONDITIONS: Food Insecurity; Food Security; Education
Keywords: Supplemental Nutrition Assistance Program-Education; nutrition education intervention

STUDY DESIGN:
Intervention Model Description: Parallel-arm intervention with inactive control group and intervention group
Who Masked: Participant
Masking Description: Participants who were recruited at the same time and location were assigned to the same treatment group to prevent knowledge of different treatment groups in the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Participants who met eligibility requirements and agreed to be randomly allocated to a treatment group. The control group participants received no lessons. Control group participants received the same study assessments at the same timepoints as the intervention group. The control group participants may have had limited contact with the nutrition educators only to update contact information, to set or remind of appointments to complete study assessments, or to receive non-nutrition or non-resource management resources.
- Intervention Group (Experimental): Participants who met eligibility requirements and agreed to be randomly allocated to a treatment group.The Intervention group participants received lessons from the nutrition educators, completed the same study assessments at the same timepoints as the control group, and may have had additional interaction with the nutrition educators in accordance with normal Indiana SNAP-Ed protocol.
  Interventions: Behavioral: Indiana SNAP-Ed

INTERVENTIONS:
Behavioral: Indiana SNAP-Ed — First four Indiana SNAP-Ed nutrition education lessons served as the intervention
  Other Names: Small Steps to Health Curriculum
  Arms: Intervention Group

SUMMARY:
The goal of the study is to determine the immediate and long-term effects of SNAP-Ed on the food insecurity of the entire household, household adults, and household children. The study also aims to determine if there is a dose-response effect on food security after receiving 4 to 10 FNP lessons and if other characteristics influence the change in food security status.

DETAILED DESCRIPTION:
FNP educators, employees of Purdue University Extension, across Indiana will help facilitate the study. FNP educators have completed CITI training as a requirement for employment through Purdue University Extension. Before recruiting study participants, participating FNP educators will attend training sessions facilitated by the co-investigators of the study. The training sessions will include instructions on how to interact with participants, answer questions related to the study, and protocol for administering surveys, keeping participant information private, and the use of identification numbers. The study goals and hypothesis will not be shared with the FNP educators in order to keep their work with the participants as unbiased as possible.

After completion of the screening survey and consent process, FNP educators will randomize participants into one of two groups: control or experimental. The FNP educators will be assigned a random number using Excel and then listed in order from least to greatest according to their random number. The first half of the FNP educators will assign their first recruited participants to the experimental group. After the first assignment, they will alternate assigning participants to either study group every other appointment. The second half of the FNP educators will assign first recruited participants to the control group. After the first assignment, they will also alternate assigning participants to either study group every other appointment. The control group will wait 1 year before starting FNP lessons. The experimental group will start FNP lessons immediately. Participants in the experimental group must take at least the first 4 FNP lessons within a time period of 4 to 10 weeks. The FNP includes 12 lessons and participants may take the additional 6 lessons if desired.

All participants will complete three 45 minute surveys. The first survey will be administered upon enrollment in the study. Participants in the experimental group will take the second survey after they have completed the first 4 lessons between 4 and 10 weeks after enrollment in the study. Control participants will take the second survey after 4 to 10 weeks with no lessons. Since participants will be recruited on a rolling basis, they will take surveys at different times within a designated time period. The third survey will be administered to both groups after 1 year of participation in the study. The third survey will be offered online. Surveys are comprised of the US Household Food Security Survey Module from the United States Department of Agriculture Economic Research Service, questions querying household and individual level characteristics, and the Indiana Food and Nutrition Program Evaluation Tool.

Two study Facebook pages will be used to keep participants engaged in the study over the year. One page will be only for the control group and another page will be only for the experimental group. Both Facebook pages will be identical in content and will prevent the experimental groups from sharing any nutrition or resource management information with the control group. The Facebook pages will include a study logo, non-nutrition and non-resource management related educational material that will cover topics such as parenting, safety, child development, fun activities to do with children, and relationships The Facebook pages will serve to keep participants engaged and to help prevent attrition. The Facebook pages will be updated monthly with new material and postings.

Researchers plan to track which study participants participate in the study Facebook pages without matching their names to their participant identification numbers. In order to carry out this procedure, researchers will make a list of all of the names that appear on the study Facebook pages at the end of recruitment in January 2014. Then researchers will send the entire list of Facebook study participants to the FNP Educators who are the only study personnel with information linking participant names to their identification numbers. FNP Educators will look through the list to see which of their clients are participating in the study and on a study Facebook page. FNP Educators will then send the researchers only the participant identification numbers of those study participants using the study Facebook page. No names matched with identification numbers will be sent to the researchers in order to preserve the privacy of the study participants through confidentiality. The purpose of collecting information on which study participants participate on the study Facebook pages will be useful for controlling for the potential confounding that exposure to the Facebook page may introduce. The Facebook pages are useful to keep participants engaged, however, they also introduce a new exposure besides the exposure of interest, the SNAP-Ed lessons. There may be differential participation in the Facebook page among the intervention and control groups and adjusting for this exposure in the analysis will allow the researchers a clearer picture of the relationship between the intervention (SNAP-Ed lessons) and the outcome of interest (food insecurity).

FNP Educators will collect electronic mailing (e-mail) addresses from all study participants willing to provide this information. The purpose of collecting e-mail addresses is to provide researchers with the ability to administer the final survey online. There is the possibility that FNP Educators will not be able to administer Survey 3 one year from administering the first survey due to a lapse in appropriations to SNAP-Ed.

ELIGIBILITY:
Inclusion Criteria:

* an interest in taking SNAP-Ed lessons
* willingness to wait 1 year to start FNP lessons
* eligibility for SNAP
* age of at least 18 years
* at least 1 child under 18 years old must live in the household
* the household located in Indiana
* ability speak and read English
* willingness to complete three 45 minute surveys at the designated time intervals
* willingness to stay in touch with research staff through a study Facebook page
* no previous participation in FNP lessons within the last year

Exclusion Criteria:

* not meeting the inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 575 (Actual)
Dates: Start 2013-09-21 (Actual); Primary Completion 2015-03-10 (Actual); Study Completion 2015-03-10 (Actual)

PRIMARY OUTCOMES:
Change in Household Food Security, Food Security Among Adults, Food Security Among Children from baseline to 1-year follow-up | Baseline assessments were completed upon recruitment and 1-year follow-up assessments were completed approximately 1 year after baseline assessments; 12-month reference period at baseline and 1-year follow-up assessments
  Score and Status as measured by 18-item US Household Food Security Survey Module at baseline and 1-year follow-up assessment time points

SECONDARY OUTCOMES:
Change in Household Food Security, Food Security Among Adults, Food Security Among Children from baseline to Post-intervention | Post-intervention food security score was assessed 4-10 weeks after baseline and included a 30-day reference period at post-intervention assessment
  Score and Status as measured by 18-item US Household Food Security Survey Module at baseline and post-intervention assessment time points

CONTACTS AND LOCATIONS:
Overall Officials: Heather A Eicher-Miller, PhD, Principal Investigator — Purdue University
Locations (1):
- Purdue University, West Lafayette, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rivera RL, Maulding MK, Abbott AR, Craig BA, Eicher-Miller HA. SNAP-Ed (Supplemental Nutrition Assistance Program-Education) Increases Long-Term Food Security among Indiana Households with Children in a Randomized Controlled Study. J Nutr. 2016 Nov;146(11):2375-2382. doi: 10.3945/jn.116.231373. Epub 2016 Sep 28. PMID 27683869
- [Background] Rivera RL, Dunne J, Maulding MK, Wang Q, Savaiano DA, Nickols-Richardson SM, Eicher-Miller HA. Exploring the association of urban or rural county status and environmental, nutrition- and lifestyle-related resources with the efficacy of SNAP-Ed (Supplemental Nutrition Assistance Program-Education) to improve food security. Public Health Nutr. 2018 Apr;21(5):957-966. doi: 10.1017/S1368980017003391. Epub 2017 Dec 4. PMID 29199629